CLINICAL TRIAL: NCT01661556
Title: Double Blind Randomized Study of 2% Miconazol Versus 4% Hydroquinone in the Treatment for Melasma.
Brief Title: Clinical Trial of Hydroquinone Versus Miconazol in Melasma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo-Cazares, Clinical Professor. Dermatology department., Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MICHQ
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Melasma
Keywords: Melasma, miconazole, hydroquinone
MeSH Terms: conditions — Melanosis | interventions — Miconazole; Clotrimazole; hydroquinone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Miconazole (Experimental): OTC topical prescription used for fungal treatment that can be useful to the treatment of melasma due to its depigmenting properties.
  Interventions: Drug: Miconazole
- Hydroquinone (Active Comparator): Hydroquinone 4% cream (Topical use) a depigmenting agent used as reference will be used as control. It will be applied twice a day for 9 weeks.
  Interventions: Drug: Hydroquinone
- Placebo (Placebo Comparator): Moisturizer cream without pharmacological effects will be used as a control.

INTERVENTIONS:
Drug: Miconazole — Miconazole 2% cream will be applied twice a day for 9 weeks. The affected surface will be washed and dried before application with a thin layer of the emulsion as indicated on the affected areas of the face.
  Other Names: Canesten; Monistat; Micatin
  Arms: Miconazole
Drug: Hydroquinone — Hydroquinone 4% cream (Topical use), will be applied twice a day for 9 weeks. The affected surface will be washed and dried before application with a thin layer of the emulsion on affected areas of the face.
  Other Names: Eldoquin; Melanex
  Arms: Hydroquinone

SUMMARY:
Melasma is an acquired discoloration of the skin characterized by brown colour changes commonly on the face.The duration of this double-blind clinical trial will be 12 weeks. The control group will receive treatment with topical Hydroquinone (4%), and the other group topical miconazole. Miconazol has antimelanotic properties and can be used as treatment for melasma patients. The estimated number of subjects to be recruited and randomized for the study is at least 30. The purpose of this study is determine if there is a difference in the effectiveness of these two agents. Melasma Area and Severity Index (MASI) score will be assessed at the beginning of the study and at weeks 4, 8, and 12. Photographs, colorimetry and histological assessment will be also evaluated. Occurrence of adverse effects will also be recorded.

DETAILED DESCRIPTION:
Melasma is a common acquired hypermelanosis in dark skin populations, usually characterized by symmetrical, irregular macules occurring in photo-exposed areas such as face. Treatment with depigmenting compounds such as hydroquinone, are still the gold standard in this condition. Miconazol has depigmented properties that could be used as part of the treatment in melasma patients. This effect is exerted by inhibiting the tyrosinase enzyme. So, the primary objective of this study is to compare the depigmenting activity of miconazole against hydroquinone.

Patients who are included in the study will be randomly assigned to receive one of the treatments, which should use for 12 weeks. The medications should be applied in the affected regions twice a day.

The evaluation of clinical improvement will be done in a blinded modality by means of the MASI score, the Global Physician Assessment, as well as colorimetry and histological melanin content. Evaluations will be held on visits at 4, 8 and 12 weeks. Skin biopsy will be taken at onset and at 12 weeks.

At the end of the study, data will be compared concerning the former parameters. All side effects will be recorded and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Mexican women over 18 years of age
* Dermatologic diagnostic of melasma
* Phototype III or more

Exclusion Criteria:

* Pregnant or breastfeeding
* Postbirth, abortion in the past 6 months
* Having an endocrine or autoimmune disease
* Under hormonal therapy of any kind including contraceptives or it´s use in the past 6 months
* Currently under treatment for melasma including sunblock
* Currently under radiation therapy, chemotherapy, immunosuppressants of any kind or phototherapy or it´s use in the past 6 months
* Having used or are consuming photosensitizing substances, oral or topical

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2015-02 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Depigmentation of melasma lesions by Colorimetry | 12 weeks
  Quantification of the colour change in the melasma lesions by means of the L axis of the CIE system. 0 is pure white, 100 y total dark.

SECONDARY OUTCOMES:
Global Physician Assessment | 12 weeks
  Clinical improvement is assessed by means of digital photographic registration (frontal, right, and left views). An independent observer clinically graded the global improvement as poor (0-25%), mild (26-50%), good (51-75%), and excellent (>75%).
MASI (Melasma Area Severity Index) | 12 weeks
  The total score would range from 0-24, involving the forehead (30%), right malar (30%), left malar (30%) and chin (10%), and using area of involvement (0=absent, 1=<10%, 2=10%-29%, 3=30%-49%, 4=50%-69%, 5=70%-89% and 6=90%-100%) and darkness (0=absent, 1=slight, 2=mild, 3=marked and 4=severe). Computation would be as follows: 0.3 A(f) D(f) + 0.3 A(lm) D(lm) + 0.3 A(rm) D(rm) + 0.1 A(c) D(c).
Melanin content by Fontana Masson stain | 12 weeks
  The Fontana-Masson Stain is specific for melanin, this histochemical reaction reveals accumulations of black material wherever melanin is located. A skin biopsy of lesions will be taken initially and at the end of study. The melanin content will be quantified by a software image analysis of the slides.

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Castanedo-Cazares, M.D., Study Director — Hospital Central "Dr. Ignacio Morones Prieto". UASLP; Amalia Reyes-Herrera, M.D., Principal Investigator — Hospital Central "Dr. Ignacio Morones Prieto". UASLP; Bertha Torres-Alvarez, M.D., Study Chair — Hospital Central "Dr. Ignacio Morones Prieto". UASLP
Locations (1):
- Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Navarrete-Solis J, Castanedo-Cazares JP, Torres-Alvarez B, Oros-Ovalle C, Fuentes-Ahumada C, Gonzalez FJ, Martinez-Ramirez JD, Moncada B. A Double-Blind, Randomized Clinical Trial of Niacinamide 4% versus Hydroquinone 4% in the Treatment of Melasma. Dermatol Res Pract. 2011;2011:379173. doi: 10.1155/2011/379173. Epub 2011 Jul 21. PMID 21822427
- [Background] Torres-Alvarez B, Mesa-Garza IG, Castanedo-Cazares JP, Fuentes-Ahumada C, Oros-Ovalle C, Navarrete-Solis J, Moncada B. Histochemical and immunohistochemical study in melasma: evidence of damage in the basal membrane. Am J Dermatopathol. 2011 May;33(3):291-5. doi: 10.1097/DAD.0b013e3181ef2d45. PMID 21317614
- [Background] Moncada B, Sahagun-Sanchez LK, Torres-Alvarez B, Castanedo-Cazares JP, Martinez-Ramirez JD, Gonzalez FJ. Molecular structure and concentration of melanin in the stratum corneum of patients with melasma. Photodermatol Photoimmunol Photomed. 2009 Jun;25(3):159-60. doi: 10.1111/j.1600-0781.2009.00425.x. PMID 19438997
- [Background] Hernandez-Barrera R, Torres-Alvarez B, Castanedo-Cazares JP, Oros-Ovalle C, Moncada B. Solar elastosis and presence of mast cells as key features in the pathogenesis of melasma. Clin Exp Dermatol. 2008 May;33(3):305-8. doi: 10.1111/j.1365-2230.2008.02724.x. PMID 18419607
- [Background] Espinal-Perez LE, Moncada B, Castanedo-Cazares JP. A double-blind randomized trial of 5% ascorbic acid vs. 4% hydroquinone in melasma. Int J Dermatol. 2004 Aug;43(8):604-7. doi: 10.1111/j.1365-4632.2004.02134.x. PMID 15304189